CLINICAL TRIAL: NCT06302608
Title: Clinical Trial on the Safety and Effectiveness of Subretinal Injection of NGGT001 for Treating Crystalline Retinal Degeneration
Brief Title: Safety and Efficacy Study of NGGT001 in Bietti Crystalline Corneoretinal Dystrophy
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xiamen Ophthalmology Center Affiliated to Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NGGT-BCD-P-2203
Record Dates: First submitted 2024-02-18; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Bietti's Crystalline Dystrophy
MeSH Terms: conditions — Bietti Crystalline Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose level 1 (Experimental): Dose level 1 will be administered
  Interventions: Genetic: NGGT001
- Dose level 2 (Experimental): Dose level 2 will be administered
  Interventions: Genetic: NGGT001

INTERVENTIONS:
Genetic: NGGT001 — Safety and Effectiveness of subretinal injection of NGGT001 for treating crystalline retinal degeneration

SUMMARY:
Evaluate the safety and tolerability of NGGT001 subretinal injection for the treatment of crystalline retinal degeneration (BCD)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Gender unlimited.
3. Diagnosed as crystalline retinal degeneration (BCD).
4. Molecular diagnosis confirms CYP4V2 mutation.
5. The best corrected visual acuity is less than 20/60.
6. Agree to take contraceptive measures within 1 year from the start of the study until administration.
7. Voluntarily sign an informed consent form.

Exclusion Criteria:

1. Insufficient number of photoreceptor cells in the retina, such as retinal thickness less than 100 μ m. Or no atrophy or pigmentation in the posterior pole area<3- Retinal disc.
2. The presence of choroidal neovascularization or other eye lesions caused by BCD, which researchers believe may affect surgical procedures or interfere with the interpretation of clinical endpoints.
3. The use of therapeutic drugs within the first 6 months of enrollment may affect experimental observation, such as Lucentis, Avastin, Conbercept, Triamcinolone acetonide, steroids, etc;
4. The treatment eye has undergone intraocular surgery, such as PDT, vitrectomy, periocular vascular bypass surgery, etc., or requires intraocular surgery during clinical research, such as cataract surgery, retinal laser therapy, etc;
5. Used or may use systemic medications that may cause eye damage, such as psoralen, tamoxifen, etc;
6. Highly sensitive or allergic to the ingredients in the experimental drug (with a history of allergies to two or more drugs or foods);
7. Abnormal and clinically significant physical examination, vital signs, laboratory tests (such as blood routine, urine routine, blood biochemistry, coagulation function, immunological tests, etc.), or abnormal indicators deemed clinically significant by researchers;
8. There are diseases or medical histories that may affect drug safety or internal processes, especially cardiovascular, liver, kidney, endocrine, digestive, lung, neurological, hematological, tumor, immune or metabolic disorders that researchers consider clinically significant.
9. Participated in clinical trials of other drugs or medical devices within 3 months prior to enrollment;
10. Female patients during pregnancy or lactation;
11. Other researchers believe that it is not suitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-05-29 (Estimated); Study Completion 2028-05-29 (Estimated)

PRIMARY OUTCOMES:
BCVA | 1 year
  ETDRS visual acuity
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 1 year
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Li, Principal Investigator — Xiamen Ophthalmology Center Affiliated to Xiamen University
Locations (1):
- Xiuju Chen, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Liu X, Cui S, Wang G, Liu Y, Qu G, Jiang L, Liu Y, Li X. Safety and Vision Outcomes Following Gene Therapy for Bietti Crystalline Dystrophy: A Nonrandomized Clinical Trial. JAMA Ophthalmol. 2025 Feb 1;143(2):126-133. doi: 10.1001/jamaophthalmol.2024.5619. PMID 39786763